CLINICAL TRIAL: NCT03957473
Title: CHEETAH: A Prospective, Multicenter Study to Evaluate the Safety and Performance of the CAT RX Aspiration Catheter in Patients With a High Thrombus Burden Acute Coronary Vessel Occlusion
Brief Title: Study of the CAT RX Aspiration Catheter When Used in Patients With Large Occlusive Thrombus in Coronary Arteries
Status: Completed | Type: Observational
Sponsor: Penumbra Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLP 15298
Record Dates: First submitted 2019-05-17; First posted 2019-05-21 (Actual); Results first posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-01

CONDITIONS: Coronary Vessel Occlusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Single Arm: Single Arm - Use of Indigo Aspiration System with CAT RX Aspiration Catheter (mechanical thrombectomy) in high thrombus burden acute coronary vessel occlusions
  Interventions: Device: Indigo Aspiration System

INTERVENTIONS:
Device: Indigo Aspiration System — Indigo Aspiration System with CAT RX Aspiration Catheter and optional Indigo Separator 4

SUMMARY:
The objective of this study is to demonstrate the safety and performance of the Indigo Aspiration System using the CAT RX aspiration catheter in a population presenting with acute high thrombus burden coronary vessel occlusion who are referred for Percutaneous Coronary Intervention (PCI).

ELIGIBILITY:
Inclusion Criteria:

* Patient age ≥ 18 years
* Patient presents to treating facility within 12 hours of symptom onset
* High thrombus burden at coronary angiography, defined as TIMI thrombus grade 4 or 5 by physician visual estimate after the guidewire crosses the target lesion
* Frontline treatment with the Indigo® Aspiration System using the CAT RX Aspiration Catheter, prior to standard of care PCI
* Target lesion is located in a native coronary artery
* Informed consent is obtained from either patient or legally authorized representative (LAR)

Exclusion Criteria:

* New onset of stroke symptoms and NIHSS > 2, prior to index procedure
* Treatment with fibrinolytic therapy for index coronary vessel occlusion
* Life expectancy less than 6 months due to any comorbidities
* Patient is unwilling or unable to comply with protocol follow up schedule and/or based on the Investigator's judgment the patient is not a good study candidate
* Participation in another investigational drug or device study that may confound the results of this study. Studies requiring extended follow-up for products that were investigational but have since become commercially available are not considered investigational studies.
* Patient is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: High thrombus burden patients presenting with acute coronary vessel occlusion who are referred for standard of care (SOC) PCI
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2019-08-22 (Actual); Primary Completion 2021-01-18 (Actual); Study Completion 2021-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: S. Jay Mathews, MD, Principal Investigator — Manatee Memorial Hospital
Locations (25):
- United States (25):
  - Cedars Sinai Medical Center, Los Angeles, California
  - St. Joseph Hospital - Orange, Orange, California
  - UCSD Medical Center, San Diego, California
  - Manatee Memorial Hospital, Bradenton, Florida
  - Clearwater Cardiovascular Consultants, Clearwater, Florida
  - Largo Medical Center, Largo, Florida
  - AdventHealth Tampa (Florida Hospital Tampa), Tampa, Florida
  - Mercy Medical Des Moines, Des Moines, Iowa
  - Jewish Hospital, Louisville, Kentucky
  - St. John Hospital, Detroit, Michigan
  - Metro Health Hospital, Grand Rapids, Michigan
  - Metropolitan Heart & Vascular, Coon Rapids, Minnesota
  - Washington University, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Desert Springs Hospital, Las Vegas, Nevada
  - University at Buffalo Medical Center, Buffalo, New York
  - NYU Langone, New York, New York
  - NC Heart & Vascular Research, Raleigh, North Carolina
  - Mercy West Hospital, Cincinnati, Ohio
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - Turkey Creek Medical Center, Knoxville, Tennessee
  - Kingwood Medical Center, Kingwood, Texas
  - Sentara Norfolk General, Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Arm
Started | 400
Completed | 370
Not Completed | 30

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 400
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 255
  >=65 years | 145
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (12.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95
  Male | 305
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14
  Not Hispanic or Latino | 378
  Unknown or Not Reported | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 12
  Native Hawaiian or Other Pacific Islander | 3
  Black or African American | 31
  White | 341
  More than one race | 1
  Unknown or Not Reported | 10
Region of Enrollment [Number; unit: participants]
  United States | 400

OUTCOME MEASURES:

1. Primary Outcome: Composite of:
Description: Cardiovascular death, recurrent myocardial infarction, cardiogenic shock, or new or worsening New York Heart Association Class IV heart failure
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 400
Participants | 14

2. Secondary Outcome: Final TIMI Flow Grade
Description: TIMI flow grading range 0-3, with higher grading representing better outcome
Time Frame: Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 400
Participants
  TIMI 0 | 0
  TIMI 1 | 0
  TIMI 2 | 10
  TIMI 3 | 390

3. Secondary Outcome: Final TIMI Thrombus Grade
Description: TIMI Thrombus grading range 0-5, with lower grading representing better outcome
Time Frame: Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 400
Participants
  Grade 0 | 398
  Grade 1 | 1
  Grade 2 | 1
  Grade 3 | 0
  Grade 4 | 0
  Grade 5 | 0

4. Secondary Outcome: Myocardial Blush Grade
Description: Myocardial blush grading range 0-3, with higher grading representing better outcome
Time Frame: Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 400
Participants
  Grade 0 | 0
  Grade 1 | 0
  Grade 2 | 1
  Grade 3 | 399

5. Secondary Outcome: Distal Embolization Rate
Time Frame: Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 400
Participants | 3

6. Secondary Outcome: Stent Thrombosis
Time Frame: 180 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 400
Participants | 9

7. Secondary Outcome: Stroke
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 400
Participants | 3

8. Secondary Outcome: Major Bleeding
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 400
Participants | 4

9. Secondary Outcome: All-Cause Mortality
Time Frame: 180 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 400
Participants | 9

10. Secondary Outcome: Cardiovascular Death
Time Frame: 180 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 400
Participants | 4

11. Secondary Outcome: Recurrent MI
Time Frame: 180 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 400
Participants | 10

12. Secondary Outcome: Cardiogenic Shock
Time Frame: 180 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 400
Participants | 8

13. Secondary Outcome: Class IV Heart Failure
Time Frame: 180 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 400
Participants | 4

14. Secondary Outcome: Incident of Device Related SAEs
Time Frame: 180 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 400
Participants | 0

ADVERSE EVENTS:
Time Frame: Procedure through 180 days
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 10/400
Serious Adverse Events (participants affected / at risk) | 144/400
Other Adverse Events (participants affected / at risk) | 30/400
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=400)
Anaemia (Blood and lymphatic system disorders) | 2
Acute myocardial infarction (Cardiac disorders) | 8
Angina pectoris (Cardiac disorders) | 5
Angina unstable (Cardiac disorders) | 5
Arteriospasm coronary (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 6
Bradycardia (Cardiac disorders) | 4
Cardiac arrest (Cardiac disorders) | 7
Cardiac failure chronic (Cardiac disorders) | 4
Cardiogenic shock (Cardiac disorders) | 3
Coronary artery disease (Cardiac disorders) | 1
Dressler's syndrome (Cardiac disorders) | 1
Ventricular arrhythmia (Cardiac disorders) | 1
Ventricular fibrillation (Cardiac disorders) | 2
Ventricular tachycardia (Cardiac disorders) | 3
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Retroperitoneal haematoma (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Chest pain (General disorders) | 5
Non-cardiac chest pain (General disorders) | 1
Vascular stent occlusion (General disorders) | 1
Vascular stent thrombosis (General disorders) | 4
COVID-19 (Infections and infestations) | 2
COVID-19 pneumonia (Infections and infestations) | 1
Osteomyelitis acute (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 6
Pneumonia influenzal (Infections and infestations) | 1
Sepsis (Infections and infestations) | 2
Septic shock (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Arterial bypass stenosis (Injury, poisoning and procedural complications) | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 3
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 2
Blood creatinine increased (Investigations) | 1
Transaminases increased (Investigations) | 1
Hypervolaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Encephalopathy (Nervous system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 7
Prescynope (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 6
Calculus urinary (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 2
Acute pulmonary eodema (Respiratory, thoracic and mediastinal disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Coronary revascularisation (Surgical and medical procedures) | 1
Accelerated hypertension (Vascular disorders) | 2
Deep vein thrombosis (Vascular disorders) | 1
Haemorrhage (Vascular disorders) | 4
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 3
Orthostatic hypotension (Vascular disorders) | 1
Coronary artery dissection (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=400)
Angina pectoris (Cardiac disorders) | 2
Arteriospasm coronary (Cardiac disorders) | 2
Atrial fibrillation (Cardiac disorders) | 2
Cardiac failure chronic (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Chest pain (General disorders) | 4
Post procedural cellulitis (Infections and infestations) | 1
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 3
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 2
Dizziness (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Haematoma (Vascular disorders) | 1
Haemodynamic instability (Vascular disorders) | 2
Haemorrhage (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-06): https://cdn.clinicaltrials.gov/large-docs/73/NCT03957473/Prot_SAP_000.pdf